CLINICAL TRIAL: NCT06749197
Title: Implementation of a Home-based Computerized Cognitive Rehabilitation Program for Patients With Acquired Brain Injury
Brief Title: Implementation of a Home-based Computerized Cognitive Rehabilitation Program for Patients With ABI
Acronym: CoRe@Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Rijndam Revalidatiecentrum (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Majanka H. Heijenbrok-Kal, PhD, Assistant professor, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13254; 10960102410036 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: cognition; cognitive impairment; attention deficit; memory disorder; computerized cognitive training; home-based training
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Attention Deficit Disorder with Hyperactivity; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cognitive training, followed by standard care (Experimental): Rehacom, standard care
  Interventions: Device: Rehacom
- Standard care, followed by cognitive training (Active Comparator): Standard care, Rehacom
  Interventions: Device: Rehacom

INTERVENTIONS:
Device: Rehacom — Home-based cognitive training program

SUMMARY:
Rationale: Patients with acquired brain injury (ABI) may suffer from persistent cognitive deficits and/or subjective cognitive complaints, especially in the domains of attention and working memory. Cognitive deficits are associated with anxiety and depression and may affect social participation and health-related quality of life (HR-QoL). Approximately 25% of the patients with ABI will be referred to an in- and/or outpatient rehabilitation center for multidisciplinary therapy to optimize recovery. Multiple studies suggest that supervised computerized cognitive training (CCT) may enhance cognitive functioning in patients with ABI. Recently, the CCT program RehaCom was introduced as an online version which is suitable for home training. In this study the feasibility and outcomes of implementing home-based CCT into a blended care pathway will be investigated in patients receiving outpatient rehabilitation therapy after ABI.

Objective: The aim of this study is to assess the feasibility and to evaluate the effect of blending a home-based CCT program (RehaCom) in standard care on cognitive functioning in patients after ABI.

The secondary aim is to evaluate the effect of this CCT program on subjective cognitive complaints, self-efficacy, psychological outcome measures and HR-QoL.

Study design: Randomized cross-over trial comparing a 5-week blended care pathway to 5 weeks of standard care within 30 patients with ABI.

Study population: Adults with ABI receiving outpatient rehabilitation therapy.

Intervention: A blended care pathway including 1 cognitive strategy training session of 1 hour per week in the outpatient rehabilitation center in combination with home-based CCT in 4 sessions of 30 minutes per week, during 5 weeks. The standard care pathway includes 2 cognitive training sessions of 1 hour per week in the outpatient rehabilitation center during 5 weeks.

Main study parameters/endpoints: Cognitive functioning (attention and working memory), self-efficacy, psychological functioning (coping, anxiety, depression) and HR-QoL, using non-invasive neuropsychological tests and standardized online questionnaires. All outcomes will be assessed at baseline (T0), after 6 weeks (T1) and after 12 weeks (T2).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the blended care pathway patients will be instructed to follow a home-based CCT program. Training at home requires a time investment from patients but will also reduce the number of visits to the rehabilitation center. Participants can choose what time of the day is most convenient for them to engage in the program in their home environment instead of traveling to the rehabilitation center for scheduled cognitive training. Increasing patients' responsibility in their recovery process may improve their self-efficacy and HRQoL.

Completion of online questionnaires also requires a certain time investment from patients and might lead to temporary fatigue. Patients may take a break at any moment and continue completing the questionnaires at a later time. By a maximum duration of 45 to 60 minutes per measurement we aim to minimize the burden for patients. There are no risks associated with participation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with acquired brain injury
* receiving outpatient rehabilitation
* sufficient command of Dutch or English language
* internet access

Exclusion Criteria:

* incapacitated patients like patients diagnosed with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
General cognition | 12 weeks
  The Montreal Cognitive Assessment (MoCA) will be used for general cognitive screening for all patients at baseline measurement and after 6 and 12 weeks.
Selective attention | 12 weeks
  The D2 test is used to measure change in visual selective attention, processing speed and concentration at the baseline visit, after 6 and 12 weeks.
Executive attention | 12 weeks
  The Stroop Test is used as a measure of mental speed, executive attention and response inhibition in all participants of the study at the baseline measurement, and after 6 and 12 weeks follow-up.
Divided attention | 12 weeks
  The Trail Making Test (TMT A&B) is used to measure change in executive function (divided attention) and processing speed at the baseline measurement, after 6 weeks and 12 weeks follow up.
Working memory | 12 weeks
  Working memory is measured in all patients at baseline measurement, after 6 weeks and at 12 weeks follow-up with the use of the Digit Span Forward (DSF) and Digit Span Backward (DSB) test (part of the Wechsler adult intelligence scale). It involves the oral presentation of spans of digits. The measure has both a 7-item digits forward task and a 7-item digits backward task, each one with its own individual score.
  Together with 'calculation' (also a part of the Wechsler adult intelligence scale), an index for working memory can be calculated.

SECONDARY OUTCOMES:
Subjective cognitive complaints | 12 weeks
  The Cognitive Failures Test (CFQ) is used for all participants at baseline measurement, after 6 weeks and at12 weeks follow-up to assess the frequency with which people experience cognitive failures in everyday life, such as absent-mindedness, slips and errors of perception, memory, and motor functioning. The total score of the scale is the sum of the ratings of the 25 individual items, yielding a score from 0-100. The CFQ has 3 sub-scales: forgetfulness, distractibility, and false triggering.
Anxiety and depression | 12 weeks
  The Dutch Hospital Anxiety and Depression Scale (HADS) is used for all participants at baseline measurement, after 6 and 12 weeks follow-up as a general measure of emotional distress and contains two sub-scales: anxiety and depression. Each sub-scale consists of 7 items, which are rated on a 0 to 3 point rating scale. Sub-scale scores ≥ 8 might indicate the presence of a depressive disorder or an anxiety disorder. Reliability and validity are adequate for several clinical populations, including multiple sclerosis and acquired brain injury.
Health-related quality of life (HR-QoL) | 12 weeks
  The EQ-5D-5L is used for all participants at baseline measurement, after 6 weeks and 12 weeks follow-up as a measurement for HR-QoL. The EQ-5D-5L consists of the 5-item EQ-5D index (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (EQ VAS). Psychometric properties of the Dutch version showed to be good. The five EQ-5D index items are summarized into one weighted overall score, which runs from 0 for the value of death to 1.00 for full health. The EQ VAS ranges from 0 to 100 (worst to best imaginable health state). For the general Dutch population average EQ-5D index = 0.843 and average EQ VAS = 81.36.
Fatigue | 12 weeks
  The Fatigue Assessment Scale (FAS) is used for all participants at baseline measurement, after 6 weeks and 12 weeks follow-up as a measurement for fatigue. The FAS is a simple and short self-administered questionnaire to assess chronic fatigue. Patients' agreement with 10 statements is rated on a 5 points Likert-scale, ranging from 1 ("never") to 5 ("always"). Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Coping | 12 weeks
  The Coping Inventory for Stressful Situations (CISS-Short Form) is used at baseline measurement, after 6 weeks and 12 weeks follow-up to measure coping styles of all participants.
  The short version of the CISS is used as a measure of coping with stressful situations. It has 21 items which are rated on a 1 to 5 point rating scale. It contains 3 subscales: task-oriented, emotion-oriented, and avoidance-oriented coping.
General Self-Efficacy | 12 weeks
  The General Self-Efficacy Scale (GSES) is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. This scale explicitly refers to personal agency, i.e., the belief that one's actions are responsible for successful outcomes. Each item is rated on a 4-point rating scale, with total scores ranging from 10 to 40. The GSES is used at baseline, after 6 and 12 weeks follow-up.

OTHER OUTCOMES:
Personality traits neuroticism and extraversion | Baseline
  The Eysenck Personality Questionnaire Brief Version (EPQ-BV) is used at baseline measurement to measure level of neuroticism and level of extraversion of all participants.
  The EPQ-BV is a revised version of the EPQ-S to measure individuals on two primary personality traits in Eysenck's personality theory (1990). It consists of two measures, one for extraversion (12 items) and one for neuroticism (12 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Rijndam Rehabilitation, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided